CLINICAL TRIAL: NCT05460390
Title: Proactive Therapeutic Drug Monitoring Based Adalimumab Therapy Optimization in Patients With Rheumatoid Arthritis
Acronym: TDM-RA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit enough participants so the study was closed.
Sponsor: Boston Medical Center (Other)
Collaborators: American Society of Health-System Pharmacists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-42873
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Therapeutic drug monitoring (TDM); Optimal trough drug concentration; Adalimumab dose optimization; Routine Assessment of Patient Index Data 3 (RAPID3)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TDM based adalimumab dose optimization group (Experimental): Therapeutic drug monitoring (TDM) provides an opportunity for a proactive and individualized therapy optimization based on serum drug concentration and anti-drug antibodies development.
  Interventions: Other: Therapeutic drug monitoring (TDM)
- Standard of care (No Intervention): Standard of care practice for RA management is based on disease activity guided therapy adjustments.

INTERVENTIONS:
Other: Therapeutic drug monitoring (TDM) — Serum trough level of adalimumab and anti-adalimumab antibody will be obtained at time of enrollment and every 3 months until the end of the study. Adalimumab dose optimization goal will be to achieve trough drug level in the range of 5 -8 μg/mL.
  Arms: TDM based adalimumab dose optimization group

SUMMARY:
Current standard of care of rheumatoid arthritis (RA) management includes a routine clinical assessment of disease activity to adjust therapy. For the most part, therapy adjustment for therapy non-response and/or suboptimal therapy response leads to therapy switch within the same class of therapy or to a different class of therapy. The lack of objective data to titrate dose of a given therapeutic agent for maximal possible efficacy makes it difficult for providers and payors to titrate dose as needed.

Therapeutic drug monitoring (TDM) provides objective data for a proactive and individualized therapy optimization based on serum drug levels and the presence or absence of anti-drug antibodies. Maintaining optimal trough drug concentration is a proven concept of therapeutics. With respect to adalimumab, this approach helps to maximize therapeutic efficacy and prevent anti-adalimumab antibody development. However, lack of drug and disease state specific published data creates a barrier for a wider adoption of TDM into clinical practice.

The objective of this single site, open label, randomized, parallel group pilot study is to investigate whether proactive therapeutic drug monitoring based adalimumab dose optimization results in higher rate of achieving and/or maintaining therapeutic goal compared to standard of care in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis
* Starting or already being treated with standard dose adalimumab, 40 mg subcutaneously (SQ) every two weeks
* Good medication adherence rate defined as Proportion of Days Covered (PDC) 80% and above

Exclusion Criteria:

* Detectable anti-adalimumab antibodies
* Overlapping immune mediated diseases
* Steroid therapy for more than 2 months prior to study enrollment
* Poor medication adherence rate (PDC < 80%)
* History of recurrent infection resulting in therapy pause
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
3 months change in proportion of patients with RA who achieve and maintain remission or low disease activity | baseline, 3 months
  Remission and low disease activity is defined as a Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) score of <2.6 and 2.6 -3.2 respectively. A DAS-28 reduction by 0.6 represents a moderate improvement, while a reduction more than 1.2 represents a major improvement.
6 months change in proportion of patients with RA who achieve and maintain remission or low disease activity | baseline, 6 months
  Remission and low disease activity is defined as a Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) score of <2.6 and 2.6 -3.2 respectively. A DAS-28 reduction by 0.6 represents a moderate improvement, while a reduction more than 1.2 represents a major improvement.
9 months change in proportion of patients with RA who achieve and maintain remission or low disease activity | baseline, 9 months
  Remission and low disease activity is defined as a Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) score of <2.6 and 2.6 -3.2 respectively. A DAS-28 reduction by 0.6 represents a moderate improvement, while a reduction more than 1.2 represents a major improvement.
12 months change in proportion of patients with RA who achieve and maintain remission or low disease activity | baseline, 12 months
  Remission and low disease activity is defined as a Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) score of <2.6 and 2.6 -3.2 respectively. A DAS-28 reduction by 0.6 represents a moderate improvement, while a reduction more than 1.2 represents a major improvement.

SECONDARY OUTCOMES:
Percent of participants who achieved low or near remission disease severity | baseline, 3 months, 6 months, 12 months
  This will be assessed with the Routine Assessment of Patient Index Data 3 (RAPID3) which is a composite disease activity index consisting of the 3 Patient Reported Outcomes, disability, pain, and patient global assessment of disease activity. Scores can range from 0 to 30 and low or near remission disease severity is defined as patients with RAPID3 disease severity score of 3.1-6 and ≤3 respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Amanuel Kehasse, PharmD, PhD, Principal Investigator — Boston Medical Center, Pharmacy
Locations (1):
- Boston Medical Center, Rheumatology Clinic, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No